CLINICAL TRIAL: NCT03583593
Title: Evaluation of Nutritional Supplement DIAMEL® Combined With Insulin in Diabetic Foot Ulcer
Brief Title: Evaluation of DIAMEL® Combined With Insulin in Diabetic Foot Ulcer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DIAMEL-DIABETICFOOT
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Diabetes Mellitus, Type 2
Keywords: Diabetes; Insulin; Diabetic Foot; Nutritional supplement; Diamel
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: It is a double blind study, that is, neither the researcher nor the patient knows if he takes placebo or the active tablet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIAMEL (Experimental): Study group that receives the active product.
  Interventions: Dietary Supplement: DIAMEL
- Placebo (Placebo Comparator): Control group receiving double-blind placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DIAMEL — Diamel is administered 6 capsules a day divided into three doses that are ingested before each meal.
  Arms: DIAMEL
Dietary Supplement: Placebo — Placebo is administered 6 capsules a day divided into three doses that are ingested before each meal.
  Arms: Placebo

SUMMARY:
Diabetic foot syndrome is one of the most frequent complications in type 2 diabetic patients. The present work is carried out with the objective of evaluating the use of DIamel combined with insulin in diabetic foot ulcers. Method. Phase II clinical trial. A study group was created that receives the active product and another control group that receives a placebo. Double-blind study with a monthly follow-up for the first 6 months and then quarterly until the end of 1 year. Complementary tests are performed every 6 months to evaluate metabolic, lipid and renal function control.

ELIGIBILITY:
Inclusion Criteria:

* Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (% B) and insulin sensitivity (% S), as percentages of a normal reference population

Exclusion Criteria:

* Manifestation of hypersensitivity to any component of the product
* Uncooperative patients
* Severe infection
* Debilitating diseases
* Steroid treatment
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Time of healing | 1 year
  The most important outcome measure is to evaluate the early healing of diabetic foot ulcers with the shape and improvements of the foot ulcers.

SECONDARY OUTCOMES:
Glycemic control | 1 year
  Glucose measures with blood test
Lipidic control | 1 year
  Triglycerides and cholesterol levels with blood test
Body mass control | 1 year
  Body mass test
Renal function control | 1 year
  Renal function measures by Creatinine Clearance Blood Test
Insulin control | 1 year
  Insulin levels measured by the Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B) and insulin sensitivity (%S), as percentages of a normal reference population

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Endocrinology, Vedado, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR